CLINICAL TRIAL: NCT03832491
Title: Effect of Game Based Approach on Oxygenation, Functional Capacity and Quality of Life in Primary Ciliary Dyskinesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Hazal Sonbahar Ulu, MSc, PT, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-180026
Record Dates: First submitted 2019-01-01; First posted 2019-02-06 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Primary Ciliary Dyskinesia; Kartagener Syndrome; Immotile Cilia Syndrome
Keywords: Primary Ciliary Dyskinesia; Kartegener Syndrome; Immotile Cilia Syndrome; Pulmonary Rehabilitation; Airway Clearance Techniques; Exergame
MeSH Terms: conditions — Ciliary Motility Disorders; Kartagener Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): Home Based Therapy: 16 patients with PCD
  Airway clearence techniques, everday of the week, during eight weeks
  Interventions: Other: Home based therapy
- Game and home based therapy group (Experimental): Game based approach programme: 16 patients with PCD
  Game based approach programme will be done using the exergame with the game console, fourty minutes three times per week for eight weeks.
  Exergame includes five games selected from two kinects games CD. Each game will be played for five games set.
  Airway clearence techniques, everday of the week, during eight weeks
  Interventions: Other: Game and home based therapy

INTERVENTIONS:
Other: Home based therapy — Airway clearence techniques
  Arms: Control Group
Other: Game and home based therapy — Game based approach programme and airway clearence techniques
  Arms: Game and home based therapy group

SUMMARY:
Impaired pulmonary function, decreased physical activity, functional capacity and depending on these factors are reported in patients with primary ciliary dyskinesia in recent studies. The purpose of this study to evaluate the effects of game based approach on pulmonary function, functional capacity and quality of life in patients with primary ciliary dykinesia.

DETAILED DESCRIPTION:
Primary ciliary dyskinesia (PCD) is an autosomal recessive hereditary disorder characterized by congenital structural abnormalities and impairment of respiratory function. Mucociliary clearance is affected by disorders in the structure and movement of cilia. That causes repeated infections in the upper and lower respiratory tract.In addition to mucociliary effects and impaired lung function, it is thought that there may be a decrease in respiratory muscle strength and functional capacity. One of the factors affecting functional capacity is the level of physical activity. For these reasons, the management of the respiratory system in patients with PCD is very important. In addition to airway clearence techniques, approaches to increase physical activity are also important. It was thought that severe physical activity could be an important determinant of cardiopulmonary functional capacity in patients with mild to moderate PCD. The level of physical activity is known to be associated with quality of life.

In literature no study investigated the effects of game based approach on oxygenation, functional capacity and quality of life in patients with PCD. Game based approach is a new method lead to increase physical activity. In literature there is no study investigated the effects of game based approach on oxygenation, functional capacity and quality of life in patients with PCD.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with PCD
* Being clinically stable
* Between 6-18 years old
* Volunteer to participate in research

Exclusion Criteria:

* Not having a stable clinical condition
* Patients with severe neuromuscular, musculoskeletal and rheumatological problems
* Patients with loss of balance
* Not being cooperative

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Functional capacity using six minute walk test | Change from baseline distance of six minute walk test in 8 weeks
  Six minute walk test will be performed in a long, straight, enclosed corridor 30 meters in length. Patients are required to walk in their walking speed with standardized instructions.
Distance of six minute walk test | Change from baseline distance of six minute walk test in 8 weeks
  The distance walked will be recorded as meters at the end of 6 minute walk test.

SECONDARY OUTCOMES:
Demographic features-Age | Before and after 8 weeks
  The age will be recorded in years.
Demographic features-Weight | Before and after 8 weeks
  Weight will be recorded in kilograms.
Demographic features-Lenght | Before and after 8 weeks
  The length will be saved in meters.
Demographic features-Body Mass Index | Before and after 8 weeks
  Body mass index will be calculated by dividing the weight by the square of the height (kg/m^2).
Vital Signs-Heart Rate | Before and after 8 weeks
  Heart rate will be recorded before and after six minute walk test, shuttle walk test, glittre ADL test, playing seated game and kinect games. The number of heart beats per minute will be evaluated before and after the tests to measure how much it has changed in 8 weeks.
Vital Signs-Systolic Blood Pressure | Before and after 8 weeks
  Systolic blood pressure will be measued before and after six minute walk test, shuttle walk test, glittre ADL test, playing seated games and kinect games. The systolic blood pressure will be evaluated before and after the tests to measure how much it has changed in 8 weeks.
Vital Signs-Diastolic Blood Pressure | Before and after 8 weeks
  Diastolic blood pressure will be measued before and after six minute walk test, shuttle walk test, glittre ADL test, playing seated games and kinect games. The diastolic blood pressure will be evaluated before and after the tests to measure how much it has changed in 8 weeks.
Vital Signs-Respiratory Rate | Before and after 8 weeks
  Respiratory rate will be recorded before and after six minute walk test, shuttle walk test, glittre ADL test, playing seated games and kinect games. The respiratory rate will be evaluated before and after the tests to measure how much it has changed in 8 weeks.
Vital Signs-Perception of dyspnea | Before and after 8 weeks
  Perception of dyspnea will be evaluated by the OMNI scale before and after six minute walk test, shuttle walk test, glittre ADL test, playing seated games and kinect games. OMNI is a perceived exertion scale as BORG perceived exertion scale. The term OMNI is an acronym for the word omnibus. This perceived exertion scale includes numerical categories from 0 to 10. The numbers on the scale show a range of exertion levels from extremely easy (0) to extremely hard (10). The perception of dyspnea will be evaluated before and after the tests to measure how much it has changed in 8 weeks.
Perception of general fatigue | Before and after 8 weeks
  Perception of fatigue will be assessed by the OMNI scale before and after six minute walk test, shuttle walk test, glittre ADL test, playing seated games and kinect games.OMNI is a perceived exertion scale as BORG perceived exertion scale.The term OMNI is an acronym for the word omnibus. This perceived exertion scale includes numerical categories from 0 to 10. The numbers on the scale show a range of exertion levels from extremely easy (0) to extremely hard (10). The perception of general fatigue will be evaluated before and after the tests to measure how much it has changed in 8 weeks.
Perception of quadriceps fatigue | Before and after 8 weeks
  Perception of quadriceps fatigue will be assessed by the OMNI scale before and after six minute walk test, shuttle walk test, glittre ADL test,playing seated games and kinect games. OMNI scale is a perceived exertion scale as BORG scale. The term OMNI is an acronym for the word omnibus. This perceived exertion scale includes numerical categories from 0 to 10. The numbers on the scale show a range of exertion levels from extremely easy (0) to extremely hard (10). The perception of quadriceps fatigue will be evaluated before and after the tests to measure how much it has changed in 8 weeks.
Pulmonary function | Before and after 8 weeks
  Pulmonary function assessed by the spirometer
Respiratory muscle strength | Before and after 8 weeks
  Respiratory muscle strength will be evaluated by the intraoral pressure measurement device.
Peripheral muscle strength | Before and after 8 weeks
  Peripheral muscle strength will be assessed by the hand held dynamometer.
Statical Balance | Before and after 8 weeks
  Statical balance will ve assessed by the flamingo balance test. The test evaluates the postural balance.In this test, a metal or wooden beam with a length of 50 cm, a height of 4 cm and a width of 3 cm is used. During this test, the participant tries to stand with a single foot in a manner similar to the flamingo position for as long as possible on the long axis of the beam. The stopwatch starts with the command. When the balance is distorted, the time is stopped and the time progresses until the next equilibrium loss.
Loss of balance of Flamingo Balance Test | Before and after 8 weeks
  Balance disturbances within 1 min are counted. If there is more than 15 loss of balance within the first 30s, the test is terminated and zero score is given.
Dynamic Balance | Before and after 8 weeks
  Dynamic balance will be evaluated by the Y balance test. The test extends to the directions determined by the lower limb of the participant and assesses the stability and stability of the participant on the other.In the test setup, 3 pieces of tape measure will be glued to the floor in an angle of 120 degrees. At the intersection of these 3 scales, one will be asked to stand on one foot with the other foot in 3 directions as anterior, posteromedial and posterolateral. At this time, the participant's balance, not to stand on the foot of the heel of the feet to stand up and extend the finger tips of the feet will be careful to touch slightly. At the end of each test, the participant will be asked to bring his foot to the side of his foot without losing the balance and touching the floor. This application will be repeated 3 times for each test.
Extending distance in Y Balance Test | Before and after 8 weeks
  Extending distance will be recorded as centimeter (cm).
Subjective Physical Activity | Before and after 8 weeks
  Subjective physical activity will ve assessed by the Bouchard Three-Day Physical Activity Questionnaire. It queries the individual's level of physical activity on weekdays and at the weekend.
Daily energy consumption in the Bouchard Three-Day Physical Activity Questionnare | Before and after 8 weeks
  The average energy calculation in kilocalories per kilogram at intervals of fifteen minutes is used to calculate daily energy consumption.
Objective Physical Activity | Before and after 8 weeks
  The objective physical activity will be evaluated by the SenseWear Armband which has three-axis accelerometer sensors during the Glittre Activity of Daily Living Test. Energy consumption will be calculated as metabolic equivalent of task (MET).
Energy expenditure while playing seated games. | Before and after 8 weeks
  Energy expenditure will be evaluated by Sense Wear Armband while playing seated games.
Energy expenditure while playing each kinect games. | Week one and half
  Energy expenditure will be assessed by Sense Wear Armband before starting to play each kinect games to determine how much energy consumption level of the games has reached during the session.
Activity of Daily Living | Before and after 8 weeks
  Activity of daily living will ve evaluated by the Glittre Activity of DailyLiving (ADL) test. Glittre ADL test is a test that provides standardized functional status assessment including activities similar to daily living activities.
Oxygenation using wearable lactate measuring instrument (BSX insight device) during Incremental Shuttle Walk Test. | Before and after 8 weeks
  1. The device is a portable NIRS LED device used to determine lactate level during the movement. BSX is housed in a compression sleeve and fitted over the gastrocnemius muscle.
Oxygenation using wearable lactate measuring instrument (BSX insight device) during Glittre Activity of Daily Living Test. | Before and after 8 weeks
  1. The device is a portable NIRS LED device used to determine lactate level during the movement. BSX is housed in a compression sleeve and fitted over the gastrocnemius muscle.
Exercise capacity using incremental shuttle walk test. | Before and after 8 weeks
  Incremental shuttle walk test will be performed in a enclosed corridor. Patients are required to turn around two cones placed 9 meters apart making the shuttle distance 10 meters long. Patients will follow the rhythm dictated by the audio signal
Quality of daily living using disease specific questioannare-Version2 (QOL-PCDV2) | Before and after 8 weeks
  The Turkish version of QOL-PCD will be used. The questionnare evaluate physical, social and emotional status in different age groups (pediatrics, adolescents, adults and parents).The total numbers of items in the questionnaires are 35 questions for parents' , 32 questions for children, 38 questions for adolescents, 40 questions for adults.

CONTACTS AND LOCATIONS:
Overall Officials: Hazal Sonbahar Ulu, MSc, PT, Principal Investigator — Hacettepe University; Deniz Inal Ince, Prof. Dr., Study Chair — Hacettepe University; Hayriye Ugur Ozcelik, Prof. Dr., Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sonbahar-Ulu H, Inal-Ince D, Saglam M, Cakmak A, Vardar-Yagli N, Calik-Kutukcu E, Sumer E, Ozcelik U. Active video gaming in primary ciliary dyskinesia: a randomized controlled trial. Eur J Pediatr. 2022 Aug;181(8):2891-2900. doi: 10.1007/s00431-022-04490-z. Epub 2022 May 10. PMID 35536410